CLINICAL TRIAL: NCT00361998
Title: Nitrofurantoin Macrocrystals 3 Days Vs. 7 Days in the Treatment of Women With Uncomplicated Cystitis
Brief Title: Nitrofurantoin Macrocrystals 3 Days Versus 7 Days in the Treatment of Women With Uncomplicated Cystitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment failed
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Clalit Health Services (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0706
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2007-03

CONDITIONS: Cystitis
Keywords: Uncomplicated Cystitis; Nitrofurantoin Macrocrystals
MeSH Terms: conditions — Cystitis | interventions — Nitrofurantoin

INTERVENTIONS:
Drug: NITROFURANTOIN MACROCRYSTALS

SUMMARY:
Our guidelines in the community recommend the use of NM for the treatment of women with community acquired UTI. While the length of treatment for uncomplicated cystitis with quinolones or TMP-SMX is three days, NM is recommended for seven days. However, there are not sufficient papers that establish the optimal length of treatment with NM in this population. The aim of this proposal is to evaluate and compare NM 3 day vs. 7 day treatment for the treatment of women with uncomplicated UTI.

DETAILED DESCRIPTION:
The aim of this proposal is to evaluate and compare NM 3 day vs. 7 day treatment for the treatment of women with uncomplicated UTI. Our design is to enroll 400 women with uncomplicated cystitis and divided according to a double-blind randomization in two groups (3 days vs. 7 days). The women will be followed 7 days and 28 days clinically and bacteriologically.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal healthy women
2. Uncomplicated cystitis

Exclusion Criteria:

1. Postmenopausal women
2. Complicated UTI
3. Women with catheter
4. Women with recurrent UTI
5. Pregnancy
6. Diabetes Mellitus

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400
Dates: Start 2006-09; Study Completion 2007-01

PRIMARY OUTCOMES:
Microbiological efficacy

SECONDARY OUTCOMES:
Clinical efficacy and side effects

CONTACTS AND LOCATIONS:
Overall Officials: Raul Raz, M.D., Principal Investigator — Infectious Diseases Unit, HaEmek Medical Center, Afula, Israel; Uzi Milman, M.D., Principal Investigator — Research Unit, Clalit Health Services, Haifa and Western-Galilee District, Israel.
Locations (1):
- Research Unit, Clalit Health Services, Haifa and Western Galillee District, Haifa, Israel